CLINICAL TRIAL: NCT01038440
Title: Evaluation of the Relationships of Time and Dose of Eicosapentaenoic Acid and Stearidonic Acid to the Changes in Eicosapentaenoic Acid Levels in Red Blood Cells
Brief Title: Time and Dose Evaluation of Stearidonic Acid (SDA) to Eicosapentaenoic Acid (EPA) in Red Blood Cells
Acronym: NK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solae, LLC (Industry)
Collaborators: Provident Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRV-09005
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Sudden Cardiac Death; Sudden Cardiac Arrest; Cardiovascular Disease
Keywords: Omega 3 fatty acids; Omega 3 Index; Stearidonic acid (SDA); Eicosapentaenoic acid (EPA); Red blood cells; Lipids; Inflammation markers
MeSH Terms: conditions — Death, Sudden, Cardiac; Cardiovascular Diseases | interventions — Safflower Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Safflower Oil
- EPA 0.5 g/d (Active Comparator)
  Interventions: Dietary Supplement: EPA
- EPA 1.5 g/d (Active Comparator)
  Interventions: Dietary Supplement: EPA
- EPA 3.0 g/d (Active Comparator)
  Interventions: Dietary Supplement: EPA
- SDA 0.5 g/d (Experimental)
  Interventions: Dietary Supplement: SDA
- SDA 1.5 g/d (Experimental)
  Interventions: Dietary Supplement: SDA
- SDA 3.0 g/d (Experimental)
  Interventions: Dietary Supplement: SDA
- SDA 6.0 g/d (Experimental)
  Interventions: Dietary Supplement: SDA

INTERVENTIONS:
Dietary Supplement: Safflower Oil — One softgel consumed daily with food
  Arms: Control
Dietary Supplement: EPA — Three different doses of EPA (0.5, 1.5 and 3.0 g/d) consumed with food daily.Subjects consuming more than 1 softgel/day (as in the groups with 1.5 and 3.0 g/d) are instructed to consume the softgels in 2 or 3 separate servings.
  Arms: EPA 0.5 g/d; EPA 1.5 g/d; EPA 3.0 g/d
Dietary Supplement: SDA — Four different doses of SDA (0.5, 1.5, 3.0 and 6.0 g/d) consumed with food daily.Subjects consuming more than 1 softgel/day (as in the groups with 1.5 and 3.0 g/d) are instructed to consume the softgels in 2 or 3 separate servings.
  Arms: SDA 0.5 g/d; SDA 1.5 g/d; SDA 3.0 g/d; SDA 6.0 g/d

SUMMARY:
The purpose of this study is to assess the relationships between dose and time of consumption of stearidonic acid (SDA) and eicosapentaenoic acid (EPA) on EPA enrichment of red blood cell (RBC) membranes in men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 21 to 65 years of age, inclusive.
2. Body mass index (BMI) 18.00-39.99 kg/m2, at visit 1 (week -2).
3. Subject is willing to avoid alcohol consumption for 24 hr prior to every clinic visit.
4. The subject has no plans to change smoking habits during the study period.
5. Subject is willing to maintain a stable body weight, current activity level, and dietary habits except for use of the study products as directed.
6. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject has coronary heart disease or a coronary heart disease risk equivalent including any of the following:

* Diabetes mellitus (or fasting glucose ≥126 mg/dL at visit 1).
* Clinical signs of atherosclerosis including peripheral arterial disease, abdominal aortic aneurysm, or certain types of carotid artery disease.
* Presence of multiple risk factors that give a person a greater than 20% chance for developing coronary artery disease within 10 years as determined by the Framingham risk index calculated at visit 1.

  2. Triglycerides ≥400 mg/dL at visit 1 (week -2). 3. If a smoker, subject smokes no more than 1 pack of cigarettes (20 cigarettes) per day.

  4. Abnormal laboratory test results of clinical importance, including, but not limited to, fasting creatinine ≥1.5 mg/dL, ALT or AST ≥1.5X the upper limit of normal or fasting glucose ≥126 mg/dL at visit 1.

  5. Uncontrolled hypertension, defined as resting systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg at screening.

  6. Use of any lipid-altering drugs, including statins, bile acid sequestrants, cholesterol absorption inhibitors, fibrates, or prescription formulations of niacin within four weeks of visit 1 and throughout the study. 7. Use of EPA/DHA from a drug or supplement within four months of visit 1 and throughout the study period.

  8. Frequent use of any non-study-related EPA/DHA containing enriched foods (such as DHA-enriched eggs) within four months of visit 1 and throughout the study period.

  9. Use of flaxseed, perilla seed, hemp, spirulina, walnut, mustard seed or black currant oil for more than one week duration within four weeks of visit 1 .

  10. Consumption of fatty fish (salmon, herring, mackerel, albacore tuna, or sardines) more than twice per month within four months of visit 1 and throughout the study period.

  11. Use of any dietary supplement known to alter lipid metabolism. 12. Use of any weight-loss medication (prescription or over-the counter) within four weeks prior to visit 1 and throughout the study.

  13. Use of any weight loss supplement or program within four weeks of visit 1 and throughout the study.

  14. Females who are pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to the use of a medically approved form of contraception throughout the study period.

  15. History or presence of significant, renal, hepatic, gastrointestinal, pulmonary, biliary, neurological or endocrine disorders.

  16. History or presence of cancer, except for non-melanoma skin cancers . 17. Current or recent history of (within 12 months of visit 1, week -1) or strong potential for alcohol or substance abuse.

  18. Use of any investigational drug within 30 days prior to visit 1. 19. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

  20. Medications and/or supplements known to influence lipid metabolism or body weight are not allowed within four weeks of visit 1. Unstable use of antihypertensive or thyroid medication will also not be permitted.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable will be the end of treatment EPA level in RBC membranes, expressed as a percent of total RBC membrane fatty acids. | 12 weeks

SECONDARY OUTCOMES:
Secondary outcome variables will include end of treatment values for: omega-3 Index (EPA + DHA as a percent of total RBC membrane fatty acids), triglycerides (TG), selected inflammatory markers | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ratna Mukherjea, PhD, Principal Investigator — Solae, LLC

REFERENCES:
- See also: Final Manuscript — http://www.ncbi.nlm.nih.gov/pubmed/22064208